CLINICAL TRIAL: NCT02558101
Title: Randomised Controlled Trial to Test Novel Invitation Methods and Materials Targeted to Increase Informed Uptake of Lung Cancer Screening in Individuals at High Risk of Lung Cancer
Brief Title: Lung Screen Uptake Trial
Acronym: Lung-SCREEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: University College London Hospitals (Other); Homerton University Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 15/0204
Record Dates: First submitted 2015-09-17; First posted 2015-09-23 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Lung Cancer
Keywords: Screening; Early detection; Health inequality; Uptake
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control invitation materials (Active Comparator): Invitation materials and strategy mimicking those of existing UK screening programmes for other cancer types
  Interventions: Behavioral: Control invitation materials
- Intervention invitation materials (Experimental): A targeted, stepped and low information burden invitation strategy and materials, specifically designed to improve uptake by reducing barriers to participation among smokers from socioeconomically deprived backgrounds.
  Interventions: Behavioral: Intervention invitation materials

INTERVENTIONS:
Behavioral: Control invitation materials — In the absence of usual care screening invitation materials, the control invitation materials and strategy are based upon the best available materials and methods of existing cancer screening programmes. These are comprised of the following:
  1. a pre-invitation letter notifying patients of the lung health check service and an information booklet mimicking those of existing screening programmes
  2. an invitation letter with a pre-scheduled appointment plus the same information booklet
  3. a reminder re-invitation letter for those who miss their appointment without cancelling
  Arms: Control invitation materials
Behavioral: Intervention invitation materials — The intervention invitation strategy is comprised of the same stages of invitation materials as the control group. The two differences are i) Instead of the information booklet they will received a targeted leaflet, and ii) the invitation and reminder letters will use indirect phrasing to explain that smokers and ex-smokers are being invited. Together, these manipulations aim to deliver a targeted, stepped and low burden approach to information provision prior to the appointment.
  Arms: Intervention invitation materials

SUMMARY:
This study tests the impact of a novel invitation strategy on attendance rates to a pre-lung cancer screening lung health check appointment. Patients will be individually randomised (1:1) to receive either control invitation materials or intervention invitation materials. Those who attend will undergo a "lung health check" and be invited to a baseline screening scan if eligibility criteria are fulfilled.

DETAILED DESCRIPTION:
Lung cancer screening using low dose computed tomography (LDCT) scans has been shown to reduce lung cancer-specific and all-cause mortality in a large United States (US) trial, and screening is now being carried out in the US. Studies have shown that participation rates are invariably low, particularly by current smokers and those from socioeconomically deprived backgrounds; groups within which high risk candidates are overrepresented.

In this study the investigators aim to improve informed participation in screening and reduce socioeconomic and smoking-related biases in participation. The investigators will identify individuals at high risk of lung cancer; specifically adults aged 60-75 who are current or recent former smokers. Eligible individuals will be invited by their General Practitioner to a "lung health check appointment" via one of two randomly allocated invitation strategies. The control materials will be similar to those used by UK screening programmes for other cancer types. The intervention materials have been designed to reduce barriers to participation among smokers from low socioeconomic status backgrounds.

Those that attend will have a lung cancer risk assessment, and if confirmed to be eligible, will undergo a baseline LDCT scan. Data will be collected with respect to demographics, risk and various clinical and radiological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Recorded as a current smoker during the year 2010 or in subsequent years since then.

Exclusion Criteria:

* Active diagnosis of lung cancer or metastases
* CT thorax within the past year
* Inability to consent to study
* Palliative care register
* GPs alert to co-morbidity that contraindicates screening or treatment for lung cancer

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1997 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2017-07-07 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Attendance to pre-allocated Lung Health Check Appointment | At an expected average of 1 year from the start of the study.
  Invitation to participation in the screening pilot will take place in blocks by GP practice and occur from day 1 until the end of recruitment (an estimated one year from the start of the study).

SECONDARY OUTCOMES:
Demographics of all those invited. | At an expected average of 1 year from the start of the study.
  Demographics of those invited to the screening pilot will take place in blocks by GP practice and occur from day 1 until the end of recruitment (an estimated one year from the start of the study).
Smoking data of those attending. | At an expected average of 1 year from the start of the study.
  This data will be recorded on enrolment of the participant to the study which will take place from 5 weeks after the start of the study until the end of recruitment (an estimated one year from the start of the study).
Data on lung cancer risk of those attending. | At an expected average of 1 year from the start of the study.
  This data will be recorded on enrolment of the participant to the study which will take place from 5 weeks after the start of the study until the end of recruitment (an estimated one year from the start of the study).
Smoking data, data on lung cancer risk, symptom history and proportion of those attending that are eligible for screening. | At an expected average of 1 year from the start of the study.
  This data will be recorded on enrolment of the participant to the study which will take place from 5 weeks after the start of the study until the end of recruitment (an estimated one year from the start of the study).
Past medical and symptom history of those attending. | At an expected average of 1 year from the start of the study.
  This data will be recorded on enrolment of the participant to the study which will take place from 5 weeks after the start of the study until the end of recruitment (an estimated one year from the start of the study).
Proportion of those invited eligible for screening. | At an expected average of 1 year from the start of the study.
  This data will be recorded on enrolment of the participant to the study which will take place from 5 weeks after the start of the study until the end of recruitment (an estimated one year from the start of the study).
Uptake of CT scans and willingness to be screening | At an expected average of 1 year from the start of the study.
  This data will be recorded on enrolment of the participant to the study which will take place from 5 weeks after the start of the study until the end of recruitment (an estimated one year from the start of the study).
Psychological burden of screening | At an expected average of 18 months from the start of the study.
  This data will be recorded at multiple timepoints following enrolment of the participant to the study. This will therefore occur from from 5 weeks after the start of the study until the end of recruitment (an estimated one year from the start of the study).
Informed decision making | At an expected average of 18 months from the start of the study.
  This data will be recorded at multiple timepoints following enrolment of the participant to the study. This will therefore occur from from 5 weeks after the start of the study until the end of recruitment (an estimated one year from the start of the study).
Radiological and clinical outcomes of those screened | At an expected average of 2 years from the start of the study.
Numbers of investigations generated from screening | At an expected average of 2 years from the start of the study.
Costs generated from screening | At an expected average of 2 years from the start of the study.
Adverse events | At an expected average of 2 years from the start of the study.
Mortality | At an expected average of 2 years from the start of the study.

OTHER OUTCOMES:
Tissue bank of biological samples from a high risk cohort | At an expected average of 1 year from the start of the study.
  This will be collected at enrolment of the participant to the study which will take place from 5 weeks after the start of the study until the end of recruitment (an estimated one year from the start of the study).

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Janes, Principal Investigator — University College, London
Locations (1):
- University College London Hospital NHS Trust, London, England, United Kingdom

REFERENCES:
- [Background] Ruparel M, Quaife SL, Ghimire B, Dickson JL, Bhowmik A, Navani N, Baldwin DR, Duffy S, Waller J, Janes SM. Impact of a Lung Cancer Screening Information Film on Informed Decision-making: A Randomized Trial. Ann Am Thorac Soc. 2019 Jun;16(6):744-751. doi: 10.1513/AnnalsATS.201811-841OC. PMID 31082267
- [Background] Ruparel M, Quaife SL, Dickson JL, Horst C, Burke S, Taylor M, Ahmed A, Shaw P, Soo MJ, Nair A, Devaraj A, O'Dowd EL, Bhowmik A, Navani N, Sennett K, Duffy SW, Baldwin DR, Sofat R, Patel RS, Hingorani A, Janes SM. Evaluation of cardiovascular risk in a lung cancer screening cohort. Thorax. 2019 Dec;74(12):1140-1146. doi: 10.1136/thoraxjnl-2018-212812. Epub 2019 Sep 26. PMID 31558626
- [Background] Quaife SL, Ruparel M, Dickson JL, Beeken RJ, McEwen A, Baldwin DR, Bhowmik A, Navani N, Sennett K, Duffy SW, Wardle J, Waller J, Janes SM. Lung Screen Uptake Trial (LSUT): Randomized Controlled Clinical Trial Testing Targeted Invitation Materials. Am J Respir Crit Care Med. 2020 Apr 15;201(8):965-975. doi: 10.1164/rccm.201905-0946OC. PMID 31825647
- [Background] Kummer S, Waller J, Ruparel M, Cass J, Janes SM, Quaife SL. Mapping the spectrum of psychological and behavioural responses to low-dose CT lung cancer screening offered within a Lung Health Check. Health Expect. 2020 Apr;23(2):433-441. doi: 10.1111/hex.13030. Epub 2020 Jan 21. PMID 31961060
- [Background] Ruparel M, Quaife SL, Dickson JL, Horst C, Tisi S, Hall H, Taylor MN, Ahmed A, Shaw PJ, Burke S, Soo MJ, Nair A, Devaraj A, Sennett K, Hurst JR, Duffy SW, Navani N, Bhowmik A, Baldwin DR, Janes SM. Prevalence, Symptom Burden, and Underdiagnosis of Chronic Obstructive Pulmonary Disease in a Lung Cancer Screening Cohort. Ann Am Thorac Soc. 2020 Jul;17(7):869-878. doi: 10.1513/AnnalsATS.201911-857OC. PMID 32164439
- [Background] Quaife SL, Ruparel M, Beeken RJ, McEwen A, Isitt J, Nolan G, Sennett K, Baldwin DR, Duffy SW, Janes SM, Wardle J. The Lung Screen Uptake Trial (LSUT): protocol for a randomised controlled demonstration lung cancer screening pilot testing a targeted invitation strategy for high risk and 'hard-to-reach' patients. BMC Cancer. 2016 Apr 20;16:281. doi: 10.1186/s12885-016-2316-z. PMID 27098676
- [Background] Ruparel M, Quaife SL, Dickson JL, Horst C, Tisi S, Hall H, Taylor M, Ahmed A, Shaw P, Burke S, Soo MJ, Nair A, Devaraj A, Sennett K, Duffy SW, Navani N, Bhowmik A, Baldwin DR, Janes SM. Lung Screen Uptake Trial: results from a single lung cancer screening round. Thorax. 2020 Oct;75(10):908-912. doi: 10.1136/thoraxjnl-2020-214703. Epub 2020 Aug 5. PMID 32759387
- [Background] Kummer S, Waller J, Ruparel M, Duffy SW, Janes SM, Quaife SL. Psychological outcomes of low-dose CT lung cancer screening in a multisite demonstration screening pilot: the Lung Screen Uptake Trial (LSUT). Thorax. 2020 Dec;75(12):1065-1073. doi: 10.1136/thoraxjnl-2020-215054. Epub 2020 Oct 21. PMID 33087548
- [Background] Balata H, Ruparel M, O'Dowd E, Ledson M, Field JK, Duffy SW, Quaife SL, Sharman A, Janes S, Baldwin D, Booton R, Crosbie PAJ. Analysis of the baseline performance of five UK lung cancer screening programmes. Lung Cancer. 2021 Nov;161:136-140. doi: 10.1016/j.lungcan.2021.09.012. Epub 2021 Sep 20. PMID 34583222
- [Background] Tammemagi MC, Ruparel M, Tremblay A, Myers R, Mayo J, Yee J, Atkar-Khattra S, Yuan R, Cressman S, English J, Bedard E, MacEachern P, Burrowes P, Quaife SL, Marshall H, Yang I, Bowman R, Passmore L, McWilliams A, Brims F, Lim KP, Mo L, Melsom S, Saffar B, Teh M, Sheehan R, Kuok Y, Manser R, Irving L, Steinfort D, McCusker M, Pascoe D, Fogarty P, Stone E, Lam DCL, Ng MY, Vardhanabhuti V, Berg CD, Hung RJ, Janes SM, Fong K, Lam S. USPSTF2013 versus PLCOm2012 lung cancer screening eligibility criteria (International Lung Screening Trial): interim analysis of a prospective cohort study. Lancet Oncol. 2022 Jan;23(1):138-148. doi: 10.1016/S1470-2045(21)00590-8. Epub 2021 Dec 11. PMID 34902336
- [Background] Hall H, Ruparel M, Quaife SL, Dickson JL, Horst C, Tisi S, Batty J, Woznitza N, Ahmed A, Burke S, Shaw P, Soo MJ, Taylor M, Navani N, Bhowmik A, Baldwin DR, Duffy SW, Devaraj A, Nair A, Janes SM. The role of computer-assisted radiographer reporting in lung cancer screening programmes. Eur Radiol. 2022 Oct;32(10):6891-6899. doi: 10.1007/s00330-022-08824-1. Epub 2022 May 14. PMID 35567604